CLINICAL TRIAL: NCT00958139
Title: Passive Prophylaxis of Lyme Disease Using Permethrin Treated Clothes
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: After year 1, there was insufficient statistical power to detect a difference in the primary outcome measure during planned study period.
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0804M3101
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Lyme Disease
Keywords: Lyme disease; tick
MeSH Terms: conditions — Lyme Disease | interventions — Permethrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Permethrin treatment of clothing (Experimental): 0.5% permethrin sprayed one time on uniform shorts, pants, and socks
  Interventions: Other: Permethrin
- Placebo (Sham Comparator): Water sprayed on uniform shorts, pants, and socks
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Permethrin — Permethrin 0.5% treatment of clothing one time
  Arms: Permethrin treatment of clothing
Other: Placebo — water sprayed on clothing one time
  Arms: Placebo

SUMMARY:
Hypothesis: Does treatment of lower extremity clothing with permethrin prevent Lyme disease?

This is a double-blind, randomized clinical trial using permethrin treatment of clothing to prevent Lyme disease.

DETAILED DESCRIPTION:
This is a double-blind, randomized clinical trial using permethrin treatment of clothing to prevent Lyme disease.

Subjects (N=200) will be recruited from camp staff to participate in the study and screened by inclusion and exclusion criteria.Qualifying subjects will be randomized to either the treatment (N=100) or non-treatment arm (N=100).

Subjects in the treatment arm will have their scout shorts, pants, and socks sprayed with 0.5% permethrin and allowed to dry. Subjects in the non-treatment arm will have their scout shorts, pants, and socks sprayed with water and allowed to dry.

Subjects will then be followed over the summer camping season to see if they develop Lyme disease. At 70 days, all subjects will have their Lyme titers rechecked to ensure that all cases of Lyme disease were documented.

Following the 70 day visit, there will be an assessment of the final study outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Summer camp staff at Tomahawk Scout Reservation
* Works in an outdoor environment
* Sleeps in an outdoor environment (platform tent)
* Present for the entire camp season (June - August)
* Informed consent

Exclusion Criteria:

* Contraindication, allergy or previous reaction to permethrin
* Inability of subject or surrogate (e.g., parent if < 18 years of age) to provide informed consent

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2008-06; Primary Completion 2008-08 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Lyme disease | Day <=70

CONTACTS AND LOCATIONS:
Overall Officials: David R. Boulware, MD, MPH, Principal Investigator — University of Minnesota
Locations (1):
- Tomahawk Scout Camp, Rice Lake, Wisconsin, United States